CLINICAL TRIAL: NCT02076750
Title: Weekly Vitamin D3 for Treatment of Hypovitaminosis D in Children and Adolescents With Inflammatory Bowel Disease
Brief Title: Weekly Vitamin D in Pediatric IBD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Subra Kugathasan, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00061627
Record Dates: First submitted 2013-12-11; First posted 2014-03-04 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Inflammatory Bowel Diseases; Skin Pigmentation
Keywords: Inflammatory Bowel Diseases; Vitamin D; Cholecalciferol; Skin Pigmentation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Pigmentation Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (cholecalciferol) 10,000 IU per 10 kg body weight (Experimental): Vitamin D3 (cholecalciferol) will be administered orally at a dose of 10,000 IU per 10 kg body weight weekly for 6 consecutive weeks. The maximum dose will be 50,000 IU weekly for patients weighing 50 kg or greater.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Vitamin D3 (cholecalciferol) 5,000 IU per 10 kg body weight (Active Comparator): Vitamin D3 (cholecalciferol) will be administered orally at a dose of 5,000 IU per 10 kg body weight weekly for 6 consecutive weeks. The maximum dose will be 25,000 IU weekly for patients weighing 50 kg or greater.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol)

SUMMARY:
The purpose of this study is to determine whether weekly dosing of oral vitamin D3 is effective in correcting low vitamin D levels in children and adolescents with inflammatory bowel disease (also known as Crohn's disease and ulcerative colitis).

DETAILED DESCRIPTION:
The role of vitamin D in skeletal health is well established. More recently, vitamin D has been implicated in multiple other disease states and is currently a topic of much discussion in the pediatric and adult medical literature. Individuals with gastrointestinal or hepatobiliary diseases that limit the absorption of dietary vitamin D and those individuals with limited sunlight exposure or darker skin color are at risk for suboptimal vitamin D status. Recent joint guidelines from the North American and European Societies of Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN and ESPGHAN, respectively) have recommended routine surveillance and treatment for vitamin D insufficiency/deficiency in children affected by inflammatory bowel diseases (IBD), namely Crohn's disease (CD) and ulcerative colitis (UC). Current recommendations are for prolonged daily dosing of oral vitamin D, but studies in children with other chronic diseases have demonstrated the benefit of improved compliance with less frequent, higher doses of vitamin D. The primary goal of this pilot study is to establish whether weekly dosing of vitamin D can correct suboptimal vitamin D status in children with inflammatory bowel disease. A secondary goal is to evaluate whether pediatric IBD patients with darker skin respond differently to vitamin D therapy than do their lighter-skinned counterparts.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of inflammatory bowel disease made by a pediatric gastroenterologist and confirmed by histopathology
2. Serum 25-OH vitamin D level <30 ng/mL at time of enrollment.
3. Age 8-21 years
4. Weight > 20 kg
5. Parent, guardian, or subject (where applicable) able to give consent/assent

Exclusion Criteria:

1. Inability to ingest oral vitamin D3 capsules
2. Presence of known hepatobiliary disease
3. Presence of known kidney disease or history of renal stones
4. Use of systemic steroids within 60 days prior to enrollment.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline serum 25-OH vitamin D level at 8 and 12 weeks | Weeks 0, 8 and 12 of study.

SECONDARY OUTCOMES:
Change from baseline serum calcium level at 8 and 12 weeks | Weeks 0, 8 and 12 of study.
Change from baseline serum parathyroid hormone level at 8 and 12 weeks | Weeks 0, 8 and 12 of study

CONTACTS AND LOCATIONS:
Overall Officials: Subra Kugathasan, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Egleston Children's Hospital, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia

REFERENCES:
- [Background] Osunkwo I, Ziegler TR, Alvarez J, McCracken C, Cherry K, Osunkwo CE, Ofori-Acquah SF, Ghosh S, Ogunbobode A, Rhodes J, Eckman JR, Dampier C, Tangpricha V. High dose vitamin D therapy for chronic pain in children and adolescents with sickle cell disease: results of a randomized double blind pilot study. Br J Haematol. 2012 Oct;159(2):211-5. doi: 10.1111/bjh.12019. Epub 2012 Aug 28. PMID 22924607
- [Background] Pappa H, Thayu M, Sylvester F, Leonard M, Zemel B, Gordon C. Skeletal health of children and adolescents with inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2011 Jul;53(1):11-25. doi: 10.1097/MPG.0b013e31821988a3. PMID 21694532